CLINICAL TRIAL: NCT04633031
Title: The Effect of Bracing on Sagittal Balance in Scoliosis, Are we Doing the Right Thing?
Brief Title: The Effect of Bracing on Sagittal Balance in Scoliosis
Status: Withdrawn | Type: Observational
Why Stopped: never approved
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: Sxxxxx
Record Dates: First submitted 2012-10-16; First posted 2020-11-17 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Idiopathic Scoliosis
Keywords: bracing; sagittal balance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group 1: Cheneau brace
  Interventions: Device: Cheneau
- Group 2: Boston brace
  Interventions: Device: Boston

INTERVENTIONS:
Device: Boston
  Groups: Group 2
Device: Cheneau
  Groups: Group 1

SUMMARY:
The goal of the study is to analyze the influence of bracing on sagittal balance in scoliosis. In special we want to observe if there is a difference between two types of TLSO-brace, namely boston and cheneau.

Retrospective analyses of Full Spine X-rays of patients who underwent bracing-therapy in the context of scoliosis.

Different spinopelvic parameters will be analyzed: pelvic incidence, pelvic tilt, sacral slope, lumbar lordosis, spinopelvic angle, spinosacral angle, thoracal kyphosis.

Four different X-rays will be reviewed for these parameters:

1. Profile before bracing therapy
2. Profile after initiation of bracing therapy
3. Profile immediately after termination of bracing therapy
4. Profile more than 3 months after termination of brace

It concerns patients with idiopathic scoliosis (exclusion of congenital scoliosis, neuromuscular scoliosis and associated spondylolisthesis).

Goal of the study is to check if treatment with TLSO-brace has a delordosing effect on sagittal balance (decrease of lumbar lordosis).

The zero-hypothesis: TLSO causes no decrease in lumbar lordosis.

Secondary goal is to compare the effect of the BOSTON TSLO-brace and otherwise the CHENEAU TLSO-brace on spinopelvic parameters and lumbar lordosis in special.

ELIGIBILITY:
Inclusion Criteria:

* late onset idiopathic scoliosis
* non-operative indication

Exclusion Criteria:

* early onset idiopathic scoliosis
* neuromuscular scoliosis
* congenital scoliosis
* associated spondylolisthesis
* operative indication

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Female and male subjects who underwent bracing therapy for an idiopathic scoliosis
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-10 (Estimated); Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Delordosing effect of TLSO brace | 3 years

SECONDARY OUTCOMES:
Difference between Boston and Cheneau brace concerning delordosing effect | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Moens, Dr, Principal Investigator — UZ Leuven
Locations (1):
- UZ Pellenberg, Pellenberg, Belgium